CLINICAL TRIAL: NCT00009932
Title: A Phase I Study Of Fenretinide Combined With Paclitaxel And Cisplatin For The Treatment Of Refractory Solid Tumors
Brief Title: Combination Chemotherapy in Treating Patients With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: OSU-00H0186; CDR0000068425 (Registry Identifier: PDQ (Physician Data Query)); NCI-2530
Record Dates: First submitted 2001-02-02; First posted 2003-06-06 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2002-10

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Cisplatin; Fenretinide; Paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: fenretinide
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining fenretinide, paclitaxel, and cisplatin in treating patients who have solid tumors that have not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose, clinical toxicity, and recommended phase II dose of fenretinide when combined with paclitaxel and cisplatin in patients with refractory solid tumors.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine the therapeutic response to this regimen in these patients.

OUTLINE: This is a dose escalation, multicenter study of fenretinide.

Patients receive oral fenretinide twice daily on days 1-7 and paclitaxel IV over 3 hours followed by cisplatin IV over 2 hours on day 2. On day 8 of course 1, patients also receive fenretinide once in the morning. Treatment repeats every 3 weeks for a maximum of 8 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response receive 2 additional courses.

Cohorts of 3-6 patients receive escalating doses of fenretinide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven refractory solid tumor for which paclitaxel and cisplatin are reasonable therapeutic options
* No active CNS disease

  * CNS metastasis allowed if measurable disease outside of the CNS and patient completed and recovered from 1 prior course of CNS radiotherapy (if clinically indicated)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least 100,000/mm3
* Absolute neutrophil count at least 1,500/mm3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* ALT and AST no greater than 2.5 times upper limit of normal (ULN) (5 times ULN if related to liver metastases)

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No severe symptomatic cardiac disease

Other:

* No clinically significant/evident retinopathy
* No other malignancy within the past 5 years except localized nonmelanoma skin cancer or carcinoma in situ of the cervix
* No uncontrolled infection
* No other significant medical or psychiatric condition that would increase risk
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 1 month before, during, and for at least 2 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior paclitaxel, cisplatin, or fenretinide
* At least 4 weeks since other prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy to only site of measurable/evaluable disease
* No prior radiotherapy to more than 25% of bone marrow

Surgery:

* At least 2 weeks since prior therapeutic surgery and recovered

Other:

* At least 4 weeks since prior routine vitamin A of at least 10,000 IU/ day or beta carotene of at least 10 mg/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A. Otterson, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio, United States